CLINICAL TRIAL: NCT04561557
Title: An Open Label Clinical Trial to Evaluate the Safety and Efficacy of CT103A Cells for the Treatment of Relapsed/Refractory Antibody-associated Inflammatory Diseases of the Nervous System
Brief Title: Safety and Efficacy of CT103A Cells for Relapsed/Refractory Antibody-associated Inflammatory Diseases of the Nervous System
Acronym: CARTinNS
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wei Wang, Professor of Neurology, President of Tongji Hospital, Tongji Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CARTinNS
Record Dates: First submitted 2020-09-10; First posted 2020-09-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Neuromyelitis Optica Spectrum Disorder; Myasthenia Gravis; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; Idiopathic Inflammatory Myopathies; Multiple Sclerosis; Autoimmune Encephalitis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD); POEMS Syndrome
Keywords: Adoptive T Cell Therapy; Chimeric antigen receptor; B-cell maturation antigen (BCMA); Autoimmune Diseases of the Nervous System
MeSH Terms: conditions — Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Neuromyelitis Optica; Myasthenia Gravis; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Myositis; Multiple Sclerosis; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; POEMS Syndrome | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAR T cells therapy，Dose level 1: 0.5 × 10^6 CAR-T cells/Kg (Experimental): The tolerability and safety of CT103A cells will be assessed in an initial dose of 0.5×10^6 CAR-T cells/Kg and three subjects will be enrolled firstly. If no dose-limiting toxicity (DLT) occurs and at least one subject benefits from the treatment, there will be two options for the investigator based on the available data: 1) three more subjects will be enrolled in the 0.5 × 10^6 CAR-T cells/Kg group and DLT will be evaluated in a total of six subjects; 2) another three subjects will be treated with 1 × 10^6 CAR-T cells/Kg instead of 0.5 × 10^6 CAR-T cells/Kg.
  If DLT occurs in one of the first three subjects, three more subjects will be enrolled in this cohort to reach the total subjects of six.
  Interventions: Biological: CT103A cells; Drug: Cyclophosphamide and fludarabine
- CAR T cells therapy，Dose level 2: 1 × 10^6 CAR-T cells/Kg (Experimental): If neither DLT nor efficacy is shown in the first three subjects, the dose of CAR-T cells will be increased to 1 × 10^6 CAR-T cells/kg to assess DLT.
  Interventions: Biological: CT103A cells; Drug: Cyclophosphamide and fludarabine
- CAR T cells therapy，Dose level 3: 0.25 × 10^6 CAR-T cells/Kg (Experimental): If DLT occurs in two subjects, whether to test the safety and efficacy in 0.25 × 10^6 CAR-T cells/kg group will be determined by the investigator based on the initial data of efficacy, PK and PD.
  Interventions: Biological: CT103A cells; Drug: Cyclophosphamide and fludarabine

INTERVENTIONS:
Biological: CT103A cells — Subjects will undergo leukapheresis to isolate peripheral blood mononuclear cells (PBMCs) to manufacture CT103A cells, during which cyclophosphamide will be administered for the purpose of lymphocytes depletion. After lymphodepletion, subjects will receive one dose treatment with CT103A cells by intravenous (IV) infusion. The initial dose of 0.5×10^6 CAR+ T cells/kg will be infused on day 0.
Drug: Cyclophosphamide and fludarabine — Subjects will receive one 3-day cycle of lymphodepletion starting 4 days prior to CT103A infusion on Day 0.
  Subjects will be given IV infusion of cyclophosphamide 300 mg/m2/day on day -4, -3 and -2, and fludarabine 30 mg/m2 over 30 minutes administered immediately after cyclophosphamide.

SUMMARY:
Antibody-mediated inflammatory diseases of the nervous system (also known as autoimmune diseases of the nervous system) are autoimmune diseases in which autoimmune cells and immune molecules attack the nervous system as the main pathogenic mechanism. In the immune response, pathogenic antibodies acting on autoantigens of the nervous system are collectively referred to as autoantibodies of the nervous system, and antibody-mediated inflammatory diseases of the nervous system can occur in the central nervous system, peripheral nervous system, and neuromuscular junctions, and muscles. In this study, we will recruit eight kinds of autoimmune diseases of nervous system including Neuromyelitis Optica Spectrum Disorder (NMOSD), Myasthenia Gravis (MG), Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP), idiopathic inflammatory myopathyand (IIM), multiple sclerosis (MS), autoimmune encephalitis (AE), Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease (MOGAD) and POEMS Syndrome. B-cell maturation antigen (BCMA) is expressed on the surface of plasma cells, thus making it an ideal target for targeted therapies. Chimeric antigen receptor (CAR) T cells against BCMA offers another potential therapeutic option to eliminate plasma cells in patients with neurological autoimmune diseases driven by abnormal antibody who still suffer recurrent attacks from conventional treatments. In the current study, the safety and efficacy of a novel CAR-T cell therapy using CT103A cells, are evaluated in patients with relapsed/refractory antibody-mediated idiopathic inflammatory diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-75 years (including 18 and 75 years);
2. Subjects with Relapsing/refractory Antibody-mediated inflammatory diseases of the nervous system without effective treatment, including:

   1. Subjects must be diagnosed as AQP4-IgG-positive NMOSD defined by 2015 criteria of IPND NMOSD and meet the following requirements: i. At least one kind of immunosuppressant has been used for more than one year with poorly-controlled symptoms; ii. Clinical evidence of at least two relapses in the last 12 months or three relapses in the last 24 months and one relapse in the preceding 12 months before screening.
   2. Subjects with MG with positive abnormal antibody, MG-ADL total score ≥ 6 points, MGFA classification II-IV defined by 2020 MGFA diagnostic criteria and meet the following requirement: i. At least one kind of immunosuppressant for standardized treatment for more than 1 year, and have one of the following poor control conditions: 1) continuous inability to affect daily life; 2) Exacerbation of MG symptoms and/or crisis attacks still occur despite standard treatment; 3) Inability to tolerate immunosuppressive therapy ii. Requires plasma exchange or maintenance therapy with IV gamma globulin
   3. Subjects with CIDP with positive abnormal antibodies, INCAT disability scale with total score of 2-9 defined by 2021 EAN/PNS diagnostic criteria and meet the following requirement: i. Standardized use of at least one first-line therapy for more than 3 months (cortisol hormone therapy, gamma globulin or plasma exchange therapy) with poorly-controlled symptoms. ii. Inability to tolerate cortisol hormones, gamma globulin, and plasmapheresis because of side effects or other conditions
   4. Subjects were diagnosed with IIM defined by 2017 European League against Rheumatism/American Rheumatology (EULAR/ACR) conference Class criteria; At least one kind of cardiac enzymes (CK, AST, ALT, ALD, LDH) ≥1.5×ULN during the screening period, or Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) ≥6, or at least one other sign of active disease within the last 6 months: MRI, EMG, or muscle biopsy; positive serological tests for myositis-specific antibodies (MSA) or myositis-associated autoantibodies (MAA), or antinuclear antibody (ANA). and meet one of the following requirements:

   i. After at least 1 month of corticosteroid therapy and standardized use of at least one immunosuppressant/modulator (eg, azathioprine, methotrexate, mycophenolate mofetil, cyclosporine, tacrolimus, Cyclophosphamide, leflunomide, intravenous gamma globulin, etc.) for more than 3 months with poorly-controlled symptoms.

   ii. ii. Inability to tolerate the above traditional regimens due to side effects or other conditions;

   e. Subjects were diagnosed with PMS (including PPMS and SPMS) or RMS according to the 2017 revision of the McDonald diagnostic criteria；EDSS score between 2 to 7 points inclusive, at screening. Subjects with RMS should meet one of the following requirements after standard therapy: i. at least two relapses in the last two years before screening. ii. at least one relapse in the last one year before screening. iii. positive Gd-enhancing MRI in the last one year before screening.

   f. Subjects were diagnosed with POEMS syndrome according to the 2021 revised IMWG diagnostic criteria and meet all of the following requirements: i. bone marrow involvement; ii. no response to traditional regimens treatment including corticosteroid, chemotherapy, protease inhibitor or inability to tolerate the above traditional regimens; iii. Have measurable lesions (refer to the 2021 revised IMWG standard) iv. VEGF > 2 ULN; v. ECOG score ≥1; vi. ONLS score ≥1.

   g. Subjects were diagnosed with autoimmune encephalitis according to the 2016 International Diagnostic Criteria for Autoimmune Encephalitis and meet all of the following requirements: i. at least one pathogenic antibody positive; ii. previously standardized use of corticosteroid, at least one immunosuppressant/modulator, including CD20 monoclonal antibody with poorly-controlled symptoms or intolerance; iii. onset of autoimmune encephalitis within 3 months prior to screening; iv. mRS Score ≥2 or CASE score ≥4.

   h. Subjects were diagnosed with MOGAD according to the 2023 International MOGAD Diagnostic criteria and meet all of the following requirements: i. a documented positive serum MOG Ab test using a cell-based assay (CBA); ii mRS Score ≥2; iii previously standardized use of corticosteroid, at least one immunosuppressant/modulator, including CD20 monoclonal antibody with poorly-controlled symptoms or intolerance.
3. All acute toxic reactions resolved to baseline or ≤ grade 1 assessed using NCI-CTCAE v5.0 except the ones adjudicated by the investigator to pose no risks on subjects.
4. Enrolled subjects must have satisfactory organ function and laboratory findings as defined by the following:i. Blood tests: absolute neutrophil count ≥ 2×109/L (or normal lower limit set by the central lab of the institution), platelets ≥ 100 × 109/L, and hemoglobin ≥ 100 g/L; ii. Liver function: total serum bilirubin, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be ≤ 1.5x the institutional normal upper limit (ULN); iii. Kidney function: CrCl ≥ 60 ml/min/1.73m2 (according to the following Cockcroft-Gault formula); iv. Electrolytes: blood potassium ≥ 3.0 mmol/L; blood calcium ≥ 2.0 mmol/L, blood magnesium ≥ 0.5 mmol/L; v. Coagulation function: fibrinogen ≥ 1.0 g/L; APTT ≤ ULN + 10s; PT ≤ ULN + 3s.
5. Blood oxygen saturation > 91% in resting state.
6. Echocardiography suggests LVEF≥ 50%.
7. Expected life expectancy ≥ 12 weeks as assessed by the investigator.
8. After signing the informed consent form, subjects and their partners must be willing to use effective and reliable method of contraception, devices or medicines, within one year after CT103A cells infusion (excluding contraception safety periods).
9. Subjects must provide written informed consent before the study begin.

Exclusion Criteria:

1. Patients do not have adequate mononuclear cells without mobilization for CAR-T cell manufacturing.
2. History of autoimmune hemolytic disease.
3. History of solid organ transplantation.
4. Patients were treated with alemtuzumab within 6 months prior to apheresis. Patients were treated with fludarabine or cladribine within 3 months prior to apheresis.
5. Patients with Papovaviruses infection.
6. Patients have been diagnosed with malignancies in the last 2 years prior to screening except for non-melanoma skin cancer, stage I cancers with complete resection and low risk of relapse, localized prostate cancer post-treatments, biopsy-confirmed in situ cervical cancer, or squamous epithelial lesion by PAP smear.
7. Chronic and active hepatitis B (HBV), hepatitis C (HCV), Human Immunodeficiency Virus (HIV) infection, CMV or syphilis infections concurrently.
8. MG crisis was not effectively controlled within 2 weeks before enrollment.
9. Known history of primary immunodeficiency (innate or acquired).
10. Patients with severe impaired cardiac function, including but not limited to the following: unstable angina, myocardial infarction (within 6 months before enrollment), congestive heart failure (≥Grade III by NYHA), severe ventricular arrhythmia.
11. Cerebrovascular accidents, including transient ischemic attack or stroke history, occurred within 6 months before enrollment.
12. Major operation or surgical treatment caused by any reason within 4 weeks before enrollment.
13. Any serious and/or uncontrolled comorbidities which may interfere with the evaluation during the study in the opinion of the investigator
14. Previous treatments: History of thymectomy within 12 months prior to CT103A infusion;
15. History of psychoactive drug abuse and failed to withdraw, or have a history of psychiatric disorders.
16. Prone to allergies or history of serious allergy.
17. Pregnant or lactating women.
18. Patients with other conditions adjudicated by the investigator as unsuitable for enrollment.

Criteria for lymphodepletion and CAR-T cells infusion:

Before lymphocyte depletion and CAR-T cells infusion, patients are evaluated and those meeting the following criteria cannot be included:

1. Blood tests: neutrophil count < 2 × 109/L, platelet count < 50 × 10^9/L;
2. Oxygen inhalation is required to maintain blood oxygen saturation ≥ 91%;
3. Patients have the following conditions, including but not limited to: new arrhythmia cannot be controlled by drugs; hypotension requiring pressor drugs; bacterial, fungal or viral infection requiring intravenous antibiotic treatment; creatinine clearance rate < 50 ml/min ;
4. Patients require maintenance support treatment within one week to meet the criteria for lymphodepletion or CAR T cell infusion.
5. Cell infusion is delayed > 7 days after lymphodepletion for any reason;
6. Patients with other conditions adjudicated by the investigator as unsuitable for lymphodepletion or cell infusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-09-22 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Types and incidence of dose-limiting toxicity (DLT) after CT103A cells infusion | Up to 28 days post CT103A infusion
  To evaluate the DLT occurred within 28 days after CT103A infusion
Incidence and severity of AEs, including changes in vital signs, physical examination, laboratory parameters, Electrocardiograms and Echocardiograms. | Up to 2 years post CT103A infusion
  To evaluate the AEs occurred within 2 years after CT103A infusion

SECONDARY OUTCOMES:
PD-Soluble BCMA | Up to 2 years post CT103A infusion
  The changes of concentration of soluble BCMA in the peripheral blood after CT103A infusion.
PD-Pathogenic antibody | Up to 2 years post CT103A infusion
  The changes of pathogenic antibody titers in peripheral blood or cerebrospinal fluid.
PD-Nfl（MS） | Up to 2 years post CT103A infusion
  The changes of peripheral blood Neurofilament Light chain (NfL) concentration in patients with MS.
PK-VCN | Up to 15 years post CT103A infusion
  The number of BCMA CAR gene copies (VCN，copies/μg DNA) in peripheral blood and cerebrospinal fluid after administration.
PK-BCMA CAR-T cells | Up to 28 days post CT103A infusion
  The concentration of BCMA CAR T cells (cells/mL) in peripheral blood after administration was detected by flow cytometry.

OTHER OUTCOMES:
NMOSD: Annualized relapse rate (ARR) | Up to 2 years post CT103A infusion
  the number of attacks divided by observed year after CT103A cells infusion
NMOSD: Accumulated total active MRI lesions | Up to 2 years post CT103A infusion
  the number of accumulate total active MRI lesions after CT103A infusion
NMOSD: Expanded Disability Status Scale (EDSS) score | Up to 2 years post CT103A infusion
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS). It consists of 7 FS (visual FS, brainstem FS, pyramidal FS, cerebellar FS, sensory FS, bowel and bladder FS, and cerebral FS) which are used to derive EDSS score ranging from 0 (normal neurological exam) to 10 (death from MS). A negative change from baseline indicates improvement. A participant was considered to have a worsening in overall EDSS score of at least 2 if baseline EDSS score was 0, or at least 1 point if baseline EDSS score is 1 to 5, or at least 0.5 point if baseline EDSS score is 5.5 or more.
NMOSD: Modified Rankin Scale | Up to 2 years post CT103A infusion
  Modified Rankin Scale (mRS) is a profoundly valid and reliable measure of disability and is broadly utilized for assessing stroke outcomes and degree of disability. We characterized a favorable outcome as mRS ranging from zero up to two, while unfavorable outcome ranging for 3 up to 6.
NMOSD: Visual acuity | Up to 2 years post CT103A infusion
  Corrected visual acuity is determine by Snellen E chart held at a distance of 5 meters. Higher score indicates better vision.
MG: Quantitative Myasthenia Gravis Score (QMG) | Up to 2 years post CT103A infusion
  The QMG score is a 13-item scale used to quantify disease severity in myasthenia gravis. The scale measures ocular, bulbar, respiratory, and limb function, grading each finding, and ranges from 0 (no myasthenic findings) to 39 (maximal myasthenic deficits).
MG: Myasthenia Gravis Activities if Daily Living (MG-ADL) Score | Up to 2 years post CT103A infusion
  The MG-ADL is an eight-question survey of symptom severity, with each response graded from 0 (normal) to 3 (most severe). Two questions concern ocular, three oropharyngeal, one respiratory, and two extremity functions. Cumulative MG-ADL scores range from 0 to 24
CIDP: Inflammatory Neuropathy Cause and Treatment (INCAT) Score | Up to 2 years post CT103A infusion
  The INCAT score comprises two parts, the arm score and the leg score. Based on a patient's level of impairment in their arms and legs, each part is scored between 0 and 5 points, resulting in an INCAT total score between 0 and 10.
CIDP: Medical Research Council (MRC) muscle function Score | Up to 2 years post CT103A infusion
  The MRC score system for testing and grading of muscle function aims to provide a standardized and objective way to assess muscle function. It ranges from 0 to 5.
CIDP: Assess changes in nerve conduction test results | Up to 2 years post CT103A infusion
  Including motor nerve distal latency, proximal latency, compound muscle motor potential (CMAP), motor nerve conduction velocity, sensory nerve conduction velocity, sural nerve potential
IMNM: Manual Muscle Testing (MMT) Score | Up to 2 years post CT103A infusion
  For MMT score, 16 muscle groups/ motions will be tested (not individual muscles). 14 of these are tested bilaterally.
IMNM: Assess the changes in serum creatine kinase levels in patients with IMNM before and after treatment. | Up to 2 years post CT103A infusion
  If the creatine kinase level drops to twice the upper limit of normal or below, it is defined as effective, and the effective rate is calculated
IMNM: Muscle MRI | Up to 2 years post CT103A infusion
  Calculating the hyperintensity of muscle MRI T2/STIR sequence in patients with IMNM
36-item Short Form Generic Health Survey (SF-36) score | Up to 2 years post CT103A infusion
  SF-36 will used to understand the health related quality-of -life of the subjects after CT103A infusion. The eight health concepts: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems; bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions will be searched. These outcomes will be grouped as physical component summary and mental component summary. The norm data is 0-100, the health related quality of life is increases as the scores are increased. The average score is 50.
EuroQol-five dimensions (EQ-SD) score | Up to 2 years post CT103A infusion
  Health status is measured with the EuroQuality of Life Five Dimensions (EQ-5D) after CT103A infusion, which includes five dimensions and is used to evaluate the quality of life of sepsis survivors. They are mobility, self-care, usual activities, discomfort or pain and depression or anxiety. Levels are coded 1-5 and a total score is then generated. Results for the demographic measured will be displayed as a percentage value.
Visual analogue scale (VAS) pain score | Up to 2 years post CT103A infusion
  usual visual analog scale (VAS) of pain is used to evaluate pain after CT103A infusion (line from 0: no pain to 10:worst pain)
Annual hospitalization rates | Up to 2 years post CT103A infusion
  The number of In-patient hospitalization is defined as a stay in hospital that goes beyond midnight of the first day of admission.
Cytokines release after CT103A infusion | Up to 2 years post CT103A infusion
  Changes of concentration( pg/mL) of cytokines ( such as ferritin, CRP, IL-6 and procalcitonin) will be analyzed after CT103A cells infusion.
Immunogenicity of CT103A cells | Up to 2 years post CT103A infusion
  Anti-drug antibodies (ADA) against CAR on CT103A cells will be analyzed after CT103A cells infusion.
Detection of RCL | Up to 2 years post CT103A infusion
  Levels of replication competent lentivirus (RCL) will be monitored after CT103A cells infusion.
Profiling of cell subtypes | Up to 2 years post CT103A infusion
  Changes in cells in infused CAR T products, blood and CSF (including proportion of CD3+ T cells, CD3+CD4+ T cells and CD3+CD8+ T cells, ratio of CD4+ T/CD8+T, and single-cell sequencing) will be analyzed after CT103A cells infusion.
MS: Annualized Relapse Rate (ARR) | Up to 2 years post CT103A infusion
  Annualized relapse rate (ARR): Number of MS relapses divided by observed year after CT103A cells infusion
MS: Time to first relapse | Up to 2 years post CT103A infusion
  Time from CT103A infusion to the first relapse of MS
MS: Number of T1 Gadolinium (Gd) | Up to 2 years post CT103A infusion
  The changes of enhancing Lesions as detected by brain Magnetic Resonance Imaging (MRI)
MS: Annualized rate of T2 lesions | Up to 2 years post CT103A infusion
  Annualized rate of T2 lesions： Number of New, and/or Enlarging T2 Hyperintense Lesions as detected by MRI divided by observed year after CT103A cells infusion
MS: Percent Change in T2 lesions volume | Up to 2 years post CT103A infusion
  The percent change of T2 lesions volume as detected by MRI from the baseline
MS: Change in EDSS | Up to 2 years post CT103A infusion
  EDSS and its associated functional system (FS) score provide a system for quantifying disability and monitoring changes in the level of disability over time. EDSS is a scale for assessing neurologic impairment in multiple sclerosis (MS).
MS: Percent of NEDA-3 | Up to 2 years post CT103A infusion
  The no evidence of disease activity-3 (NEDA-3), defined as no relapse, no disability worsening, and no MRI activity
MS: 3-month CDP | Up to 3 months post CT103A infusion
  Time to onset of 3-month CDP as assessed by EDSS score
MS: 6-month CDP | Up to 6 months post CT103A infusion
  Time to onset of 6-month CDP as assessed by EDSS score
MS: Patient Reported Outcomes (PRO) | Up to 2 years post CT103A infusion
  Including Fatigue Symptoms and Impacts Questionnaire -Relapsing Multiple Sclerosis (FSIQ-RMS), General Anxiety Disorder Scale (GAD-7), Patient Health Questionnaire (PHQ-9), Health Utilities Index (HUI-III), Multiple Sclerosis Impact Scale (MSIS-29).
POEMS syndrome: Overall Response Rate (ORR) | Up to 2 years post CT103A infusion
  Definition of Response:
  1. There is a one-point improvement in ECOG performance score; and/or
  2. ≥ 50% reduction in ONLS score.
POEMS syndrome: Hematological response rate | Up to 2 years post CT103A infusion
  Hematological response rate: Percentage of subjects who achieved partial response (PR) or better according to 2021 IMWG Uniform Response Criteria.
POEMS syndrome: Neural response rate | Up to 2 years post CT103A infusion
  Definition of Neural Response: a) There is a one-point improvement in ONLS score; and/or b) ≥ 15% reduction in mNIS+7 score.
POEMS syndrome: Change in VEGF | Up to 2 years post CT103A infusion
  The changes of VEGF levels after CT103A cells infusion.
POEMS syndrome: PET response rate | Up to 2 years post CT103A infusion
  PET response rate: Percentage of subjects who achieved response according to 2021 IMWG Uniform Response Criteria.
POEMS syndrome: Response rate of other organs | Up to 2 years post CT103A infusion
  Percentage of subjects who achieved response of other organs.
AE: Time to ≥1point improvement in modified Rankin score (mRS) | Up to 2 years post CT103A infusion
  Time to ≥1point improvement in modified Rankin score (mRS) from baseline without rescue therapy.
AE: Time to first relapse | Up to 2 years post CT103A infusion
  Time to first relapse: Time from CT103A infusion to the first relapse of AE (days).
AE: Epilepsy | Up to 2 years post CT103A infusion
  The time to seizure-free (Patients with autoimmune encephalitis have sympotmatic seizures in the acute phase) or the time from seizure-free (without rescue therapy) to rescue therapy.
AE: Change in CASE | Up to 2 years post CT103A infusion
  The changes of Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score from baseline.
AE: Change in MoCA | Up to 2 years post CT103A infusion
  The changes of Montreal Cognitive Assessment Scale (MoCA) total scores from baseline.
AE: Change in CGI | Up to 2 years post CT103A infusion
  The changes of Total Clinical Global Impressions (CGI) score from baseline.
AE: Change in GCS | Up to 2 years post CT103A infusion
  The changes of Total Glasgow Coma Score (GCS) from baseline.
AE: Change in MMSE | Up to 2 years post CT103A infusion
  The changes of Total Minimum Mental State Examination Score (MMSE) from baseline.
AE: Number of FBDS | Up to 2 years post CT103A infusion
  The number of faciobrachial dystonic seizure (FBDS) in patients with LGI1 antibody-positive encephalitis.
MOGAD: Annualized relapse rate | Up to 2 years post CT103A infusion
  Annualized recurrence rate: The number of MOGAD relapses divided by observed year after CT103A cells infusion
MOGAD: Time to first relapse | Up to 2 years post CT103A infusion
  Time to first relapse: Time from CT103A infusion to the first relapse of MOGAD.
MOGAD: MS: Number of T1 Gadolinium (Gd) | Up to 2 years post CT103A infusion
  The changes of enhancing Lesions as detected by MRI.
MOGAD: Change in EDSS | Up to 2 years post CT103A infusion
  The changes of EDSS score from baseline.
MOGAD: Change in MoCA | Up to 2 years post CT103A infusion
  The changes of MOCA score from baseline.
MOGAD: Change in MoCA | Up to 2 years post CT103A infusion
  The changes of MMSE score from baseline.
All patients: Change in mRS | Up to 2 years post CT103A infusion
  The changes of mRS score from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin C, Dong MH, Zhou LQ, Chu YH, Pang XW, He JY, Shang K, Xiao J, Zhu L, Ye H, Cai SB, Wang D, Bu BT, Meyer Zu Horste G, Li CR, Tian DS, Wang W. Anti-BCMA CAR-T therapy in patients with progressive multiple sclerosis. Cell. 2025 Nov 13;188(23):6414-6423.e11. doi: 10.1016/j.cell.2025.09.020. Epub 2025 Oct 15. PMID 41101309
- [Derived] Dong MH, Mei ZC, Zhou LQ, Heming M, Xu LL, Liu YX, Pang XW, Chu YH, Cai SB, Ye H, Shang K, Xiao J, Meyer Zu Horste G, Wang W, Qin C, Tian DS. Anti-BCMA CAR-T cell therapy in relapsed/refractory chronic inflammatory demyelinating polyneuropathy. Med. 2025 Sep 12;6(9):100704. doi: 10.1016/j.medj.2025.100704. Epub 2025 May 26. PMID 40425008
- [Derived] Keam SJ. Equecabtagene Autoleucel: First Approval. Mol Diagn Ther. 2023 Nov;27(6):781-787. doi: 10.1007/s40291-023-00673-y. Epub 2023 Sep 2. PMID 37658205